CLINICAL TRIAL: NCT05793320
Title: Prospective Histopathologic and Clinical Evaluation of Patients Undergoing Carpal Tunnel Release With Risk Markers for Amyloidosis
Brief Title: Carpal Tunnel Release With Risk Factors for Amyloidosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Interim Chairman & Medical Director, Professor of Orthopaedic Surgery, Department of Orthopaedic Surgery & Service Line, Wayne State University School of Medicine, Henry Ford Health, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16239-01
Record Dates: First submitted 2023-03-16; First posted 2023-03-31 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carpal Tunnel Release (Experimental)
  Interventions: Procedure: Carpal Tunnel Release Surgery

INTERVENTIONS:
Procedure: Carpal Tunnel Release Surgery — Carpal tunnel release surgery used to take a biopsy to diagnose amyloidosis and determine whether or not carpal tunnel syndrome can predict who's at risk for having amyloidosis.

SUMMARY:
Bilateral carpal tunnel syndrome has been demonstrated in previous literature to be a warning sign for potential amyloidosis. One study has been performed in which patients with bilateral carpal tunnel syndrome underwent tissue biopsy (either tendon sheath or transverse carpal ligament) at the time of carpal tunnel release to determine the strength of association as well as most common subtypes. However, no study has been done demonstrating whether or not patients with amyloid-positive carpal tunnel biopsy would benefit from an early referral to cardiology for a work-up of potential cardiac amyloidosis. In our study, patients with bilateral carpal tunnel symptoms who are indicated for carpal tunnel release would be identified in clinic and undergo biopsy for congo red staining at the time of surgery. All patients with positive biopsy results would be referred to cardiology. Outcomes would include the rate of amyloid positivity, common subtypes, and echocardiographic findings after cardiac referral.

ELIGIBILITY:
Inclusion Criteria:

Positive screening is defined as two characteristics from Tier 1 or one characteristic from Tier 1 and one from Tier 2 Tier 1

* Male > 50 years old
* Female > 60 years old
* Bilateral carpal tunnel symptoms or prior release surgery Tier 2
* Spinal stenosis
* History of biceps tendon rupture
* Atrial fibrillation or flutter (active or previous history)
* Pacemaker
* Congestive heart failure
* Family history of transthyretin amyloidosis (ATTR)

Exclusion Criteria:

* Unable or unwilling to follow up with cardiology.
* Previous diagnosis of cardiac amyloidosis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males older than 50 years old and females older than 60 years old are eligible.
Enrollment: 250 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-08-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Rate of amyloid positivity | Biopsy sent for testing immediately after the procedure
  How many patients who participate in study have positive biopsy for amyloidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Day, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Main Campus, Detroit, Michigan, United States